CLINICAL TRIAL: NCT00829751
Title: The Physiological Consequence of Silicone-hydrogel Care-solution Bio-incompatibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Jerry R. Paugh, OD, PhD, Professor, Associate Dean for Research, Southern California College of Optometry at Marshall B. Ketchum University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 08-8
Record Dates: First submitted 2009-01-23; First posted 2009-01-27 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Contact Lens Solution Toxicity
Keywords: staining; toxicity; fluorometry; dye diffusion; anterior chamber

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ReNu Multiplus (Active Comparator): Purevision lenses will be soaked in ReNu Multiplus
  Interventions: Device: PureVision lenses soaked in ReNu Multiplus
- OptiFree RePlenish (Active Comparator): PureVision lenses will be soaked in OptiFree RePlenish
  Interventions: Device: PureVision lenses soaked in OptiFree RePlenish

INTERVENTIONS:
Device: PureVision lenses soaked in ReNu Multiplus — Purevision silicone hydrogel lenses
  Arms: ReNu Multiplus
Device: PureVision lenses soaked in OptiFree RePlenish — Purevision silicone hydrogel lenses soaked in OptiFree RePlenish
  Arms: OptiFree RePlenish

SUMMARY:
The purpose of this study is to more objectively evaluate potential lens-material/care solution bio-incompatibilities. We will do this by measuring corneal staining and the amount of fluorescein dye diffusion into the eye.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Best correctable vision to 20/40 in each eye.
* Possess a functional spectacle prescription to allow adequate vision during the de-adaptation and fluorometry measurement period.
* No known ocular or systemic allergies, which may interfere with contact lens wear.
* No known systemic disease, or need for medication that may interfere with contact les wear (i.e. antihistamines, beta-blockers, steroids, ect.).

Exclusion Criteria:

* Subjects demonstrating any medical condition that may affect the results of this study SHOULD NOT be enrolled. The following are specific conditions that exclude subjects from enrollment in this study.
* Eye (ocular) or systemic allergies that may interfere with contact lens wear.
* Clinically significant corneal swelling (greater than 3 or 4 on a 0-4 scale), corneal blood vessel growth (vascularization), corneal staining, bulbar redness, tarsal redness, or any other abnormality of the cornea that may cause unsafe contact lens wear.
* Are taking part in any other study or have taken part in a study within the last 14 days.
* Are pregnant, or anticipating to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The level/amount of sodium fluorescein dye in the anterior chamber at post wear timepoints | On day of experiment

SECONDARY OUTCOMES:
Corneal staining level post lens wear | On day of study

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Paugh, OD, PhD, Principal Investigator — Southern California College of Optometry at Marshall B. Ketchum University
Locations (1):
- Southern California College of Optometry, Fullerton, California, United States